CLINICAL TRIAL: NCT05119322
Title: Study of the Use of a Home Test for the Detection of Gluten Immunogenic Peptides in Urine and Its Effect on Gluten-free Diet Adherence
Brief Title: Use of a Home Test for Gluten Detection in Urine and Its Effect on Gluten-free Diet Adherence
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of resources
Sponsor: Biomedal S.L. (Other)
Collaborators: FUNDACION IHP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLUTENDETECT
Record Dates: First submitted 2021-10-26; First posted 2021-11-15 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Celiac Disease; Treatment Adherence; Adolescent
Keywords: Celiac disease; Gluten-free diet adherence; Adolescent; Gluten immunogenic peptides; Urine tests
MeSH Terms: conditions — Celiac Disease; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Intervention and control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlutenDetect home urine test (Experimental): The GlutenDetect home urine test group will receive home use tests for GIP detection in urine to self-monitor the GFD. Tests will be used at their discretion, but using at least 8 tests during the study period (1/week), so that they may receive immediate qualitative feedback regarding the presence of biomarkers of gluten exposure in their urine and they will have to register the results obtained. Additionally, patients will collect a urine and a stool sample every 4 weeks to evaluate their adherence to the GFD in the laboratory.
  Interventions: Diagnostic Test: GlutenDetect home urine test
- Control group (No Intervention): The control group will not receive any home urine tests but will collect a urine and a stool sample every 4 weeks with the purpose of evaluating their adherence to the GFD in the laboratory.

INTERVENTIONS:
Diagnostic Test: GlutenDetect home urine test — GFD compliance self-asessment using a home rapid test for GIP detection in urine.
  Arms: GlutenDetect home urine test

SUMMARY:
The use of a home rapid test for the detection of gluten immunogenic peptides (GIP) in urine of treated adolescent patients with celiac disease (CD) could facilitate the adherence to the gluten-free diet (GFD) and contribute to symptoms control and quality of life improvement.

This single centre, randomized, unblinded, controlled study consists of 4 run-in weeks period followed by 8-weeks study period in which patients will be randomized to intervention group (home urine GIP testing) or the control group (no home urine GIP testing). The 12-week study will involve surveys, home stool and urine collection, home urine GIP test performance, and two study visits with the gastroenterologists.

The main outcome is to determine whether the self-monitoring of the GFD with GIP testing in urine improves adherence to the GFD in treated adolescent patients with CD (measured by CDAT-Celiac Dietary Adherence Test, GFD adherence evaluation by gastroenterologist and rates of gluten exposure in urine and/or stool measured at a central laboratory) and subsequently improves quality of life (CDDUX-Coeliac Disease Dutch Questionnaire) and reduces symptoms (CSI-Celiac Symptoms Index questionnaire).

DETAILED DESCRIPTION:
Hypothesis: the use of a home rapid test for the detection of gluten immunogenic peptides (GIP) in urine of treated adolescent patients with celiac disease (CD) could facilitate the adherence to the gluten-free diet (GFD) and contribute to symptoms control and quality of life improvement.

Objectives:

Primary objective: to determine in adolescent patients with CD whether the self-monitoring of the GFD with GIP testing in urine changes treatment adherence (intervention group) in comparison with patients that do not use the test (control group) measured by 1 - CDAT-Celiac Dietary Adherence Test; 2 - GFD adherence evaluation by gastroenterologist; 3- Detection rates of GIP in urine and/or stool (to be measured at a central laboratory); 4- Detection rates of GIP in urine (to be measured by home rapid tests).

Secondary objectives: to determine whether the use of the home test for GIP detection in urine samples of treated patients with CD leads to 1 - change of quality of life (CDDUX-Coeliac Disease Dutch Questionnaire); 2- change of symptoms (CSI-Celiac Symptoms Index questionnaire).

Study design: Single centre, randomized, unblinded, controlled, study. The study will consist of 4 run-in weeks period followed by 8-weeks study period in which patients will be randomized to intervention (home urine GIP testing) or the control group (no home urine GIP testing).

Study participants: adolescent patients with CD, diagnosed by European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) guidelines, that have been following a strict GFD for at least 2 years.

Study procedure:

1. Patient enrolment.
2. Run-in period (4 weeks): all participants will: A- complete quality of life questionnaire (CDDUX); B - complete GFD adherence questionnaire (CDAT); C - complete food diary for 4 consecutive days and GFD adherence will be evaluated by gastroenterologist; D - complete symptom questionnaire (CSI); E - be instructed in the use of the tests and sample collection; F - collect at the beginning and end of the period urine and stool samples.
3. Study weeks (8): patients will be randomized to either the control or the study group by block randomization (size 4) using WINPEPI (Programs for epidemiologists for Windows) v11.65 (Abramson, J.H.). The study group will receive home use tests for GFD monitoring to be used at their discretion (but using at least 8 tests during the study period (1/week) so that they may receive immediate qualitative feedback regarding the presence of biomarkers of gluten exposure in their urine and they will have to register the results obtained. The control group will not receive the tests. Additionally, all patients will collect a urine and a stool sample every 4 weeks with the purpose of evaluating their adherence to the GFD. All collected samples will be kept frozen until their analysis and will be brought to the centre by the patients at the end of the study. All samples will be sent to a central laboratory for their analysis (Biomedal S.L., Seville, Spain).
4. At the end of the study, patients will be evaluated as in the run-in period (post-intervention).

Number of participants: with an alpha risk of 5%, a beta risk of 20% (80% of statistical power) and an estimated rate reduction of 0.33 the sample size needed was 66 subjects (33 subjects per group). The calculation was made using the tool Calculadora de Grandària Mostral (GRANMO) v7.12 April 2012 (Municipal Institute of Medical Research, Barcelona, Spain).

Measurements: 1- Home rapid test (GlutenDetect, Biomedal S.L., Seville, Spain) for GIP determination in urine samples, laboratory rapid test (iVYCHECK GIP Urine, Biomedal S.L., Seville, Spain) for GIP determination in urine samples and ELISA test (iVYLISA GIP Stool, Biomedal S.L., Seville, Spain) for GIP determination in stool samples; 2- CD related symptoms (CSI questionnaire); 3- quality of life questionnaire (CDDUX); 4- GFD adherence questionnaire (CDAT); 5- GFD adherence evaluation by specialist (questionnaire and food diary); 6 - test results for the study group. Samples will be analysed in a central laboratory (Biomedal S.L., Seville, Spain).

Statistical analysis: Will be done with IBM SPSS Statistics 25.0 for Windows (IBM Corporation, Armonk, New York, United States). 1- Difference in all parameters between and within the control and the study groups. Results will be compared at baseline, week 4 and week 12. 2- Differences in all parameters between patients with positive GIP testing compared to those with negative GIP testing (both home and laboratory GIP measurements). 3 - number of additional tests used by the patients since they will receive 24 tests and they must perform only 8 tests. They can use the additional test at their discretion.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to take part in the study.
* Signed informed consent.
* Diagnosis of CD confirmed by biopsy and/or serology.
* Ability to: provide urine and stool samples, perform the home tests, and register results.

Exclusion Criteria:

* Not precise diagnostic of CD.
* Comorbid condition that in the opinion of the investigator would interfere with the study.
* Lack of willingness to take part in the study.
* Inability to use the test or provide samples.
* Frequent voluntary GFD transgressions.
* To provide less than 70% of the required samples.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gluten-free adherence change | 8 weeks
  Number of participants adherent to GFD in intervention and control arms as assessed by Celiac Dietary Adherence Test (CDAT), change from baseline in scores on the test after 8 weeks of intervention. The scores on the CDAT have a scale from 7 to 35. A score of <13 is considered as good diet adherence and a score >17 is considered as bad diet adherence.
Gluten-free adherence change | 8 weeks
  Number of participants adherent to GFD in intervention and control arms as assessed by GFD adherence evaluation questionnaire by gastroenterologist, change from baseline in level of diet adherence on the questionnaire after 8 weeks of intervention. The scores have a scale from 0 to 32 and social questions (5) have a yes/no answer. A score of 0-7 and "no" in all social questions is considered excellent diet adherence; a score of 8-15 and "no" in all social questions is considered good diet adherence; a score of 8-15 and "yes" in one social question is considered regular diet adherence; a score of 16-24 and "yes" in two social questions is considered regular diet adherence; a score of 16-24 and "yes" in three social questions is considered bad diet adherence; a score of 25-32 and "yes" in two social questions is considered bad diet adherence; a score of 25-32 and "yes" in three social questions is considered very bad diet adherence.
Gluten-free adherence change | 8 weeks
  Number of participants adherent to GFD in intervention and control arms as assessed by detection of GIP in urine and/or stool samples (measured at a central laboratory), change from baseline in GIP qualitative and quantitative results after 8 weeks of intervention.
Gluten-free adherence change | 8 weeks
  Number of participants adherent to GFD in intervention group as assessed by detection of GIP in urine samples (measured by home rapid tests), change from baseline in GIP qualitative results after 8 weeks of intervention.

SECONDARY OUTCOMES:
Quality of life change | 8 weeks
  Number of participants with affected quality of life in intervention and control arms as assessed by Coeliac Disease Dutch Questionnaire (CDDUX), change from baseline in scores from after 8 weeks of intervention. The scores on the CDDUX are recoded into a scale from 1 to 100. A score of 1-20 is considered very bad, 21-40 is bad, 41-60 is neutral, 61-80 is good, and 81 to 100 is very good.
Symptoms change | 8 weeks
  Number of participants with CD symptoms in intervention and control arms as assessed by Celiac Symptoms Index questionnaire (CSI), change from baseline in symptom scores after 8 weeks of intervention. The scores on the CSI are recoded into a scale from 16 to 80. A score of ≥38 is considered as symptomatic.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Coto Alonso, Principal Investigator — Biomedal S.L.; Ángel Cebolla Ramírez, Study Director — Biomedal S.L.; Joaquín Reyes Andrade, Principal Investigator — Fundación IHP
Locations (1):
- Grupo IHP, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comino I, Real A, Vivas S, Siglez MA, Caminero A, Nistal E, Casqueiro J, Rodriguez-Herrera A, Cebolla A, Sousa C. Monitoring of gluten-free diet compliance in celiac patients by assessment of gliadin 33-mer equivalent epitopes in feces. Am J Clin Nutr. 2012 Mar;95(3):670-7. doi: 10.3945/ajcn.111.026708. Epub 2012 Jan 18. PMID 22258271
- [Background] Moreno ML, Cebolla A, Munoz-Suano A, Carrillo-Carrion C, Comino I, Pizarro A, Leon F, Rodriguez-Herrera A, Sousa C. Detection of gluten immunogenic peptides in the urine of patients with coeliac disease reveals transgressions in the gluten-free diet and incomplete mucosal healing. Gut. 2017 Feb;66(2):250-257. doi: 10.1136/gutjnl-2015-310148. Epub 2015 Nov 25. PMID 26608460
- [Background] Gerasimidis K, Zafeiropoulou K, Mackinder M, Ijaz UZ, Duncan H, Buchanan E, Cardigan T, Edwards CA, McGrogan P, Russell RK. Comparison of Clinical Methods With the Faecal Gluten Immunogenic Peptide to Assess Gluten Intake in Coeliac Disease. J Pediatr Gastroenterol Nutr. 2018 Sep;67(3):356-360. doi: 10.1097/MPG.0000000000002062. PMID 29916953
- [Background] Comino I, Fernandez-Banares F, Esteve M, Ortigosa L, Castillejo G, Fambuena B, Ribes-Koninckx C, Sierra C, Rodriguez-Herrera A, Salazar JC, Caunedo A, Marugan-Miguelsanz JM, Garrote JA, Vivas S, Lo Iacono O, Nunez A, Vaquero L, Vegas AM, Crespo L, Fernandez-Salazar L, Arranz E, Jimenez-Garcia VA, Antonio Montes-Cano M, Espin B, Galera A, Valverde J, Giron FJ, Bolonio M, Millan A, Cerezo FM, Guajardo C, Alberto JR, Rosinach M, Segura V, Leon F, Marinich J, Munoz-Suano A, Romero-Gomez M, Cebolla A, Sousa C. Fecal Gluten Peptides Reveal Limitations of Serological Tests and Food Questionnaires for Monitoring Gluten-Free Diet in Celiac Disease Patients. Am J Gastroenterol. 2016 Oct;111(10):1456-1465. doi: 10.1038/ajg.2016.439. Epub 2016 Sep 20. PMID 27644734
- [Background] Costa AF, Sugai E, Temprano MP, Niveloni SI, Vazquez H, Moreno ML, Dominguez-Flores MR, Munoz-Suano A, Smecuol E, Stefanolo JP, Gonzalez AF, Cebolla-Ramirez A, Maurino E, Verdu EF, Bai JC. Gluten immunogenic peptide excretion detects dietary transgressions in treated celiac disease patients. World J Gastroenterol. 2019 Mar 21;25(11):1409-1420. doi: 10.3748/wjg.v25.i11.1409. PMID 30918433
- [Background] Comino I, Segura V, Ortigosa L, Espin B, Castillejo G, Garrote JA, Sierra C, Millan A, Ribes-Koninckx C, Roman E, Rodriguez-Herrera A, Diaz J, Silvester JA, Cebolla A, Sousa C. Prospective longitudinal study: use of faecal gluten immunogenic peptides to monitor children diagnosed with coeliac disease during transition to a gluten-free diet. Aliment Pharmacol Ther. 2019 Jun;49(12):1484-1492. doi: 10.1111/apt.15277. Epub 2019 May 10. PMID 31074004
- See also: GlutenDetect website — https://glutendetect.es/en/
- See also: iVYDAL website — https://ivydal.biomedal.com/en/professional-use-tests/